CLINICAL TRIAL: NCT01185574
Title: Vitamin D for Improving Metabolic Control and Depressive Symptoms in Women With Diabetes; The Sunshine Study
Brief Title: Vitamin D for Improving Metabolic Control and Depressive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Sue Penckofer, Professor, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201255
Record Dates: First submitted 2010-08-18; First posted 2010-08-20 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Depressive Symptoms; Diabetes
MeSH Terms: conditions — Depression; Diabetes Mellitus | interventions — Ergocalciferols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vitamin D supplementation (Experimental): The study medication (a capsule of 50,000 IU of vitamin D2) will be administered once a week for six months.
  Interventions: Dietary Supplement: Vitamin D supplementation

INTERVENTIONS:
Dietary Supplement: Vitamin D supplementation — Vitamin D2 50,000 IU will be administered once a week for six months.
  Other Names: Drisdol

SUMMARY:
This study will examine whether weekly vitamin D supplementation in women with significant depressive symptoms and diabetes will exhibit improved mood and metabolic control. If supplementation with Vitamin D is beneficial, it will be a simple and cost-effective method for treatment. Women will be targeted since they have greater depression and worse metabolic control than men with diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 and older
2. medically stable type 2 diabetes with HBA1c <9%.
3. significantly elevated depressive symptoms as measured by a score greater than or equal to 14 using the Center for Epidemiologic Studies Depression Tool (CES-D.

Exclusion Criteria:

1. vitamin D levels of 32 ng/dl or greater
2. malabsorption problems (e.g., crohn's disease, celiac sprue)
3. hypercalcemia-level greater than 10.5 mg/dl
4. Severe complications of diabetes (amputation, blindness, or renal problems) 5) Women with low thyroid function

6) active suicidal ideation, a history of bipolar depression, psychotic disorders, and current alcohol or substance disorders. Active treatment for depression (e.g., antidepressant therapy) will not be exclusion criteria 7) Any serious chronic illness that may impact on their health-related quality of life and treatment effect 8) Women who are pregnant 9) Women who have had bariatric surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Metabolic control | 6 months

SECONDARY OUTCOMES:
depressive symptoms | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States